CLINICAL TRIAL: NCT03333629
Title: Connecting the Dots: An RCT Integrating Standardized ASD Screening, High-Quality Treatment, and Long-Term Outcomes
Brief Title: Promoting Positive Outcomes for Individuals With ASD: Linking Early Detection, Treatment, and Long-term Outcomes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: University of California, Davis (Other); University of Connecticut (Other)
Responsible Party: Principal Investigator, Diana Robins, Professor, Drexel University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: R01MH115715 (NIH)
Record Dates: First submitted 2017-09-08; First posted 2017-11-07 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Autistic Disorder; Early Detection; Early Intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced early detection (Experimental): Providers will receive training to administer enhanced early detection strategies.
  Interventions: Behavioral: Enhanced early detection
- Usual care (No Intervention): Providers will not change their early detection strategies, but will be monitored.

INTERVENTIONS:
Behavioral: Enhanced early detection — standardized screening
  Arms: Enhanced early detection

SUMMARY:
Autism spectrum disorder (ASD) is defined by impaired social engagement and social communication, and repetitive, restricted, or stereotyped behaviors and interests. The average age of diagnosis in the US is after the fourth birthday. However, children who start ASD-specific early intervention have better outcomes than children start later. The current study will address a gap identified by the US Prevention Services Task Force, namely that children detected through screening respond positively to early intervention. This study will directly relate early detection strategies to early intervention, and measure the impact of age of intervention onset on outcomes when children are entering kindergarten. Local pediatric providers will be randomized to provide either usual care, or to an experimental condition in which autism early detection strategies are enhanced through the addition of specific procedures. Across all sites, 8,000 children will be recruited through their participating pediatric practice. Qualifying children will receive up to one year of early intensive behavioral intervention, after getting an ASD diagnosis. Primary outcome measures will include children's cognitive functioning and ASD symptom severity, which will be measured at multiple time points. The investigators predict that this study will inform early detection strategies which will result in improving children's social and cognitive functioning, mitigating lifespan disability, reducing societal costs, and improving personal well-being and productivity of individuals with ASD.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a serious neurodevelopmental disorder defined by impaired social engagement and social communication, in addition to the presence of repetitive, restricted, or stereotyped behaviors and interests. Although many cases of ASD can be detected when children are less than two years old, the average age of diagnosis in the US is still after the fourth birthday. However, evidence demonstrates that children who start ASD-specific early intervention have better outcomes than children who do not start treatment until later ages. In 2006 and 2007, American Academy of Pediatrics recommended three early detection approaches to improve identification of children at risk for ASD: ongoing developmental surveillance at every well-child check-up, routine broad developmental screening at three infant/toddler ages, and ASD-specific screening at two toddler ages. When these early detection strategies are used with all children attending well-child check-ups, the age of ASD detection is lower, and children who are diagnosed have the opportunity to start ASD-specific early intervention at younger ages than if they had not been detected. Yet in 2016, the US Preventive Services Task Force (USPSTF) indicated that current evidence is insufficient to recommend universal ASD screening, given the lack of experimental studies demonstrating positive outcomes for treated children that are detected through screening. The current study will address this gap. This study will directly relate early detection strategies to early intervention, and measure the impact of age of intervention onset on outcomes when children are entering kindergarten. The study will be conducted by investigators from three sites: Drexel University; the University of California, Davis; and the University of Connecticut. Local pediatric providers will be enrolled in the study, and their practices will be randomized to provide either usual care, or to an experimental condition in which autism early detection strategies are enhanced through the addition of specific procedures. Children attending well-child visits at participating practices will then be enrolled. Across all sites, 8,000 children will be recruited through their participating pediatric practice. As part of the study, qualifying children will receive up to one year of early intensive behavioral intervention, using an evidence-based manualized treatment. Primary outcome measures will include children's cognitive functioning and ASD symptom severity, which will be measured at multiple time points. Exploratory outcomes will include children's adaptive functioning, kindergarten readiness, and social reciprocity, as measured by experimental eye tracking and parent-child interaction ratings. This study also will examine the impact of the screening intervention on physician attitudes and on parent empowerment and stress. Finally, investigators will examine potential moderators of outcomes, to determine whether initial symptom severity, cognitive ability, or socioeconomic status affects children's long-term outcomes. The investigators predict that this study will inform early detection strategies which will result in improving children's social and cognitive functioning, mitigating lifespan disability, reducing societal costs, and improving personal well-being and productivity of individuals with ASD.

ELIGIBILITY:
Inclusion Criteria:

* child attended 18 m visiting at participating pediatric practice
* legal guardian is fluent in English or Spanish

Exclusion Criteria:

* child has severe sensory or motor deficit that precludes completing standardized evaluation

Ages: 16 Months to 58 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2087 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in ASD Symptom Severity | Change from pre-treatment to immediately post-treatment; 10 minutes
  ASD symptom severity will be measured with the Brief Observation of Social Communication Change (BOSCC)
Change in Cognitive Functioning | Change from pre-treatment to immediately post-treatment; 60 minutes
  Cognitive functioning will be measured by the Mullen Scales of Early Learning (MSEL).

SECONDARY OUTCOMES:
Adaptive Functioning | Immediately post-treatment, 48 m, 60 m; 45 minutes
  Vineland Adaptive Behavior Scales-3
ASD Symptoms - secondary measure1 | 48 m, 60 m; 45 minutes
  Autism Diagnostic Observation Schedule, Second Edition (ADOS-2)
Kindergarten Readiness | 60 m; 45 minutes
  Developmental Indicators for the Assessment of Learning-4
Social Engagement | Immediately post-treatment, 48 m, 60 m; 15 minutes
  Eye tracking paradigms will assess aspects of social engagement (i.e., social orienting, motivation, and cognition)
Long-term change in Cognitive Functioning | 48 m, 60 m; 60 minutes
  Cognitive functioning will be measured by the Mullen Scales of Early Learning (MSEL)
Parent-Child Social Engagement | Immediately post-treatment, 48 m, 60 m; 15 minutes
  Parent-child social engagement will be measured with the Joint Engagement Rating Inventory, which is applied to video recordings of the Communication Play Protocol.
ASD symptoms - secondary measure2 | Immediately post-treatment, 48 m, 60 m; 20 minutes
  PDD Behavior Inventory
ASD symptoms - secondary measure3 | 48 m, 60 m; 10 minutes
  BOSCC
Long-term change in Cognitive Functioning (alternative) | 48 m, 60 m; 60 minutes
  and for children who reach ceiling on the MSEL, we will use the Differential Differential Abilities Scales-II (DAS-II) will be used for children too advanced for Outcome 7

CONTACTS AND LOCATIONS:
Overall Officials: Diana Robins, PhD, Principal Investigator — Drexel University
Locations (3):
- United States (3):
  - University of California, Davis, Sacramento, California
  - University of Connecticut, Storrs, Connecticut
  - Drexel University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded to the National Database for Autism Research (NDAR) semi-annually
Time Frame: semi-annual uploads beginning December 2018
Access Criteria: as per NDAR requirements

REFERENCES:
- [Derived] Vivanti G, Algur Y, Ryan V, McClure LA, Fein D, Stahmer AC, Wieckowski AT, Robins DL. The Impact of Using Standardized Autism Screening on Referral to Specialist Evaluation for Young Children on the Autism Spectrum: A Cluster-Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2025 Jun;64(6):686-698. doi: 10.1016/j.jaac.2024.08.502. Epub 2024 Oct 15. PMID 39454668
- [Derived] McClure LA, Lee NL, Sand K, Vivanti G, Fein D, Stahmer A, Robins DL. Connecting the Dots: a cluster-randomized clinical trial integrating standardized autism spectrum disorders screening, high-quality treatment, and long-term outcomes. Trials. 2021 May 2;22(1):319. doi: 10.1186/s13063-021-05286-6. PMID 33934719